CLINICAL TRIAL: NCT00568880
Title: A Phase I/II Trial of Hydroxychloroquine Added to Bortezomib for Relapsed/Refractory Myeloma
Brief Title: Hydroxychloroquine and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01407
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydroxychloroquine Added to Bortezomib (Experimental): Dose escalated by cohorts Hydroxychloroquine 200-600 mg pill every other day. Bortezomib 1.0-1.3mg/m2 IV, days 1, 4, 8, and 11 of each 21 day cycle.
  Interventions: Drug: bortezomib; Drug: hydroxychloroquine

INTERVENTIONS:
Drug: bortezomib — bortezomib 1.0-1.3mg/m2 IV
  Other Names: Velcade
Drug: hydroxychloroquine — hydroxychloroquine 200 mg pill
  Other Names: Plaquenil

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxychloroquine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving hydroxychloroquine together with bortezomib may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of hydroxychloroquine when given together with bortezomib and to see how well it works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the dose-limiting toxicities and maximum tolerated dose of hydroxychloroquine when added to a standard-dose regimen of bortezomib for treatment of patients with relapsed or refractory multiple myeloma.

Secondary

* To obtain a preliminary estimate of the toxicity rate and response rate of this combination at the maximum tolerated dose.
* To confirm preclinical evidence showing synergistic effects of hydroxychloroquine and bortezomib by correlating response rate with blood levels of hydroxychloroquine and degree of autophagy inhibition in repeated bone marrow samples.

OUTLINE: This is a phase I dose-escalation study of hydroxychloroquine followed by a phase II study.

* Phase I: Patients receive oral hydroxychloroquine every other day for 2 weeks. Patients then receive oral hydroxychloroquine 1-3 times daily or every other day and bortezomib IV twice a week for 2 weeks. Treatment with hydroxychloroquine and bortezomib repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Once the maximum tolerated dose (MTD) for hydroxychloroquine is determined, additional patients are accrued to the phase II portion of the study.
* Phase II: Patients receive hydroxychloroquine (at the MTD determined in phase I) and bortezomib as in phase I.

Blood and bone marrow samples are collected periodically during the study for correlative studies by mass spectrometry, proteasome inhibition assays, pharmacokinetic analysis and assessment of aggresome formation, autophagy inhibition, and apoptosis by protein electrophoresis and serum free light-chain analysis.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed multiple myeloma
* Documented relapse or continued disease after at least one prior therapy (which may include autologous and allogeneic bone marrow transplantation)
* Need for further therapy for myeloma, as determined by the patient's treating physician
* Age greater than 18 years

Exclusion Criteria

* Baseline peripheral neuropathy of grade 2 or higher
* History of allergic reactions to compounds of similar chemical or biologic composition to bortezomib or hydroxychloroquine
* Prior dose-limiting toxicity with bortezomib
* Known macular degeneration or retinopathy (diabetic or otherwise), porphyria, or psoriasis. Patients with well-controlled psoriasis may participate in the study provided that they are under the care of a specialist in this condition who agrees to monitor the patient for exacerbations.
* Other conditions that would require therapy with hydroxychloroquine, including but not limited to systemic lupus, rheumatoid arthritis, porphyria cutanea tarda, and malaria treatment or prophylaxis
* ECOG performance status >2 (for definition, see section 0)
* Life expectancy of less than 3 months
* Lack of adequate organ or bone marrow function based on lab values drawn ≤ 14 days before beginning treatment.
* Concurrent treatment with a different investigational regimen. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
* Treatment with other anti-myeloma agents, including thalidomide or lenalidomide, within the 14 days prior to initiating hydroxychloroquine. Treatment with corticosteroids will be permitted up to 7 days prior to initiating hydroxychloroquine. Corticosteroids that are being used for other diseases are permitted if the dose is less than the equivalent of 20 mg of prednisone daily. Concurrent therapy with bisphosphonates through the study period is permitted at the discretion of the treating physician. Concurrent hematopoietic growth factors are also permitted, including filgrastim or pegfilgrastim, epoetin alpha, and darbepoetin alpha
* Known central nervous system involvement. The poor prognosis and progressive neurological dysfunction associated with central nervous system involvement would confound the evaluation of neurological and other adverse events. The presence of calvarial lytic lesions or plasmacytomas is not an exclusion criterion if there is no central nervous system involvement.
* Concurrent malignancy other than basal cell carcinoma of the skin, squamous cell carcinoma of the skin, any carcinoma in situ, or localized prostate adenocarcinoma (stage T1a or T1b) with a stable PSA for a period of at least 4 months. Patients with a prior malignancy treated with chemotherapy, biologic agents, and/or radiation are eligible for this study if they have completed therapy ≥4 years previously with no evidence of recurrent disease. Patients with a prior malignancy treated with surgery alone are eligible for this study if they have completed therapy ≥2 years previously with no evidence of recurrent disease.
* Uncontrolled intercurrent illness including, but not limited to: uncontrolled ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability to understand the informed consent document or unwillingness to consent. Written informed consent must be obtained from all patients before study entry.
* Pregnancy or breastfeeding.
* Unwillingness to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation for men and women of child-bearing potential.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2011-06-22 (Actual); Study Completion 2011-06-22 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Day 1 of each cycle (each cycle is 21 days)
  This is assessed using International Working Group criteria.

SECONDARY OUTCOMES:
Effects of regimen on the autophagy pathway | at baseline, prior to bortezomib on Day1 and 8 of cycle 1, prior to bortezomib on Day 1 of cycle 2 (each cycle is 21 days)
  Measure peripheral blood mononuclear cells
AV accumulation during therapy | Day 1 and 8 of the first cycle and on Day 1 of each subsequent treatment cycle (each cycle is 21 days)
  mean AVs / Bone Marrow plasma cell

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Vogl DT, Stadtmauer EA, Tan KS, Heitjan DF, Davis LE, Pontiggia L, Rangwala R, Piao S, Chang YC, Scott EC, Paul TM, Nichols CW, Porter DL, Kaplan J, Mallon G, Bradner JE, Amaravadi RK. Combined autophagy and proteasome inhibition: a phase 1 trial of hydroxychloroquine and bortezomib in patients with relapsed/refractory myeloma. Autophagy. 2014 Aug;10(8):1380-90. doi: 10.4161/auto.29264. Epub 2014 May 20. PMID 24991834